CLINICAL TRIAL: NCT03120494
Title: Evaluating the Feasibility and Acceptability of Implementing a PrEP Program in PR-CoNCRA (San Juan, Puerto Rico)- Part B
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Puerto Rico Community Network for Clinical Research on AIDS (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Puerto Rico PrEP study- Part B
Record Dates: First submitted 2017-04-11; First posted 2017-04-19 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2017-04

CONDITIONS: HIV/AIDS
Keywords: HIV prevention, high risk MSM, sero-discordant couples, PrEP
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: All subjects will receive same treatment with study drug
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects at risk of HIV (Experimental): 25 high risk MSM and 50 negative partners in a sero-discordant couple will be recruited and emtricitabine and tenofovir (Truvada) for PrEP will be provided, per guidelines, for one year
  Interventions: Drug: Emtricitabine and Tenofovir

INTERVENTIONS:
Drug: Emtricitabine and Tenofovir — All subjects will be provided study drug for use daily for one year.
  Other Names: Truvada

SUMMARY:
75 subjects at risk for HIV infection (25 high risk MSM and 50 sero-discordant couples) will be recruited. All subjects will receive Truvada for pre-exposure prophylaxis or PrEP, as well as routine medical evaluations during one year. Subjects will be managed according to CDC's guidelines on the management of PrEP as a tool for HIV prevention.

DETAILED DESCRIPTION:
75 subjects at risk for HIV infection (25 high risk MSM and 50 sero-discordant couples) will be recruited. All subjects will receive Truvada for PrEP, as well as routine medical evaluations during one year. Subjects will be managed according to CDC's guidelines on the management of PrEP as a tool for HIV prevention.

All subjects will have a total of at least 8 study visits during which routine assessment are performed for patients on Truvada for PrEP. Apart from offering routine medical care, a baseline questionnaire that includes socio-demographic variables, PrEP knowledge and acceptability and sexual conducts will be offered. At the 6 months visit, an abbreviated sexual conducts questionnaire will be offered.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male, female or transgender female age 21 or older
2. Subject provides written informed consent.
3. Subject provides written authorization for use and disclosure of protected health information (PHI).
4. Subject has one of the following risk factors:

   * male, female or transgender female or female sexual partner of an HIV-infected individual, ideally who is not virologically suppressed
   * high risk MSM as defined by: having unprotected sexual intercourse with at least two male partner in the last 6 months, or
   * diagnosed with an STI in the past 6 months
5. Baseline eCrCl of ≥60 ml/min (calculated using the CKD-EPI formula)
6. Negative Hepatitis B serology
7. No medical contraindications to the use of PrEP
8. Confirmed HIV negative by 5th generation (AB/antigen) HIV test

Exclusion Criteria:

1. younger than 21 years of age
2. unable to provide consent
3. Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice).
4. Positive pregnancy test: Women of childbearing potential must have a negative serum or urine pregnancy test within 1 week prior to study entry. Pregnancy testing will also be performed in enrolled female participants prior to any study procedures being performed
5. Baseline eCrCl <60 ml/min
6. Positive Hepatitis B serology to avoid potential flares upon product discontinuation
7. Any medical contraindication to the use of PrEP or any other conditions deemed by the study investigator to exclude the subject's participation in the study
8. HIV infected
9. Signs and symptoms of acute HIV infection
10. For sero-discordant couples: upon review of HIV positive partner's chart, evidence of resistance to any of the components of the study drug.
11. Illness or other condition that, in the opinion of the PI, may interfere with study participation at the time of enrollment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Trans-gender female will be allowed in the study
Enrollment: 75 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Retention in care | 12 months
  Retention to follow up clinical visits based on completed and missed visits
Treatment adherence | 12 months
  Determine adherence to study drug based on pill count and died blood spots (DBS)
PrEP knowledge | 12 months
  Measure the level of education of the study subjects in the topic of PrEP using a questionnaire

SECONDARY OUTCOMES:
Study drug safety | 12 months
  Determine safety of study drug based on AE reports related to treatment
Study drug safety | 12 months
  Determine safety of study drug based on safety laboratories monitoring, reported as percentage of participants with abnormal laboratory values
HIV sero-prevalence | 12 months
  Determine the sero-prevalence of the study subjects receiving PrEP based on the number of study subjects diagnosed with HIV during study duration.
Changes in sexual risk behaviors | 12 months
  Measure changes from baseline sexual risk behaviors after initiating use of study drug, specifically frequency of unprotected sexual intercourse according to sexual behaviors questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian M Tamayo-Agrait, MD, Principal Investigator — PR-CoNCRA
Locations (1):
- Puerto Rico Community Network for Clinical Research on AIDS (PR-CoNCRA), San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No